CLINICAL TRIAL: NCT00491634
Title: Phase II Trial of Fludarabine Combined With Intravenous Treosulfan and Allogeneic Hematopoietic Stem-cell Transplantation in Patients With Chemo-refractory or Previously Untreated Acute Myeloid Leukemia and Myelodysplastic Syndrome.
Brief Title: Treosulfan-based Conditioning for Transplantation in AML/MDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Avichai Shimoni MD (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Avichai Shimoni MD, Dr. Avichai Shimoni, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-07-3116-AN-CTIL
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: acute myeloid leukemia; myelodysplastic syndrome; allogeneic stem cell transplantation; reduced-intensity conditioning; treosulfan
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — treosulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): treosulfan
  Interventions: Drug: treosulfan

INTERVENTIONS:
Drug: treosulfan — 12 g/m2 x 3 days
Drug: Treosulfan — 12 g/m2 x 3

SUMMARY:
The study hypotheses is that the introduction of dose escalated treosulfan, in substitution to busulfan, will reduce toxicity after allogeneic transplantation while improving myeloablation and and disease control in patients with AML and MDS not eligible for standard transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Age less than physiologic 68 years.
2. Patients with AML and MDS not eligible for standard TBI- or Busulfan-based myeloablative conditioning due to age, concurrent medical condition, or extensive prior therapy (e.g. age > 55 years for HLA-matched sibling transplants or > 50 for matched unrelated donor transplants, prior / concomitant pulmonary, liver, or other organ complications).
3. This study will only include patients with chemo-refractory disease or previously untreated active disease.

   A. acute myeloid leukemias (AML) according to WHO classification (> 20% myeloblasts in peripheral blood or bone marrow at diagnosis) in induction failure, PR, untreated or chemo-refractory relapse. Patients must have > 10% marrow blasts at the time of transplantation.

   B. myelodysplastic syndromes (MDS) according to WHO classification (< 20% myeloblasts in peripheral blood and bone marrow at diagnosis), indicated for allogeneic transplantation:

   - refractory anaemia with excess blasts (RAEB-1 and RAEB-2) with no prior therapy
4. Patients must have an HLA matched related or unrelated donor willing to donate either peripheral blood stem cells or bone marrow. Matching is based on high-resolution class I (HLA-A, -B, -C) and class II (HLA-DRB1, -DQB1) typing. The goal is to transplant > 3 x 106 CD34+ cells per kg body weight of the recipient -

Exclusion Criteria:

1. Bilirubin > 3.0 mg/dl, transaminases > 3 times upper normal limit
2. Creatinine > 2.0 mg/dl
3. ECOG-Performance status > 2
4. Uncontrolled infection
5. Pregnancy or lactation
6. Abnormal lung diffusion capacity (DLCO < 40% predicted)
7. Severe cardiovascular disease
8. CNS disease involvement
9. Pleural effusion or ascites > 1 liter
10. Known hypersensitivity to fludarabine or treosulfan
11. Psychiatric conditions/disease that impair the ability to give informed consent or to adequately co-operate -

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
disease-free survival | 2 years after transplantation

SECONDARY OUTCOMES:
treatment-related mortality, GVHD, relapse, overall survival | 2 year after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Nagler, MD, Principal Investigator — Chaim Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Kroger N, Shimoni A, Zabelina T, Schieder H, Panse J, Ayuk F, Wolschke C, Renges H, Dahlke J, Atanackovic D, Nagler A, Zander A. Reduced-toxicity conditioning with treosulfan, fludarabine and ATG as preparative regimen for allogeneic stem cell transplantation (alloSCT) in elderly patients with secondary acute myeloid leukemia (sAML) or myelodysplastic syndrome (MDS). Bone Marrow Transplant. 2006 Feb;37(4):339-44. doi: 10.1038/sj.bmt.1705259. PMID 16415898